CLINICAL TRIAL: NCT01718522
Title: The Application and Advantage of Sensor Augmented Pump (SAP) Therapy Under Daily Conditions (Registerstudie Zur Anwendung Und Nutzen Der Sensorunterstützten Pumpentherapie (SuP) Unter Alltagsbedingungen)(RANSuP)
Brief Title: Registry of Use and Application of Sensor Augmented Pump (SAP) Therapy Under Daily Life Conditions
Acronym: RANSuP
Status: Completed | Type: Observational
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Other Study IDs: CEN_G_DB_1
Record Dates: First submitted 2012-10-17; First posted 2012-10-31 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Intervention Group: Patients treated with sensor augmented pump (SAP) therapy with insulin pump Paradigm VEO® and use continuous glucose monitoring (CGM).
  Interventions: Device: sensor augmented pump (SAP)

INTERVENTIONS:
Device: sensor augmented pump (SAP)

SUMMARY:
The purpose of this registry is to collect the real life data on Sensor Augmented pump (SAP) therapy usage in type 1 Diabetes mellitus (DM) patients treated with Medtronic Insulin pumps and continuous glucose monitoring systems in Germany.

DETAILED DESCRIPTION:
The purpose of this registry is to reflect the daily practice with Sensor Augmented Pump (SAP) therapy usage in Type 1 Diabetes Mellitus (DM) patients treated with Medtronic insulin pumps (Paradigm VEO®) and continuous glucose monitoring systems in Germany. In addition, the aim is of this registry is to support:

* obtain reimbursement for SAP therapy in Germany
* building a platform (advisory committee) for discussion of SAP data.
* looking for deficits with implementation of glucose sensor data in diabetes therapy management and development of "follow-up education" materials.

This is a national multi-center, post-market non-interventional prospective study with CE marked and commercially available devices and consumables.

The study will be conducted from March 2012 to April 2013 in Germany. The duration of individual patient participation is 3 to 6 months.

Health outcomes will be measured in approximately 75 patients between 6-65 years old diagnosed with Type 1 DM over a period of at least 3 months in approximately 15 centers. The patients are under treatment of Paradigm VEO® without any additional insulin injections and use continuous glucose monitoring, or patients that are not using continuous glucose monitoring, but that are willing to start with SAP. The enrolled subjects have a first visit inquiring the status data (including upload of device data in CareLink software, Hemoglobin A1c (HbA1c) value measurement) without any intervention. Thereafter, the SAP therapy is optimized based on individual continuous glucose monitoring (CGM) data during a second visit one month later and then a last visit like the first visit in which the status will be determined.

Parameters of glycemic control will be measured, such as the frequency of hypoglycemia (glucose values ≤ 70 mg/dl), over a period of 30 days after the first patient's visit (Visit 1) and after the visit 2 when an adjustment of the therapy has been discussed with the patient based on the collected CGM results between the two first visits.

ELIGIBILITY:
Inclusion Criteria:

* patients with signed informed consent
* Type 1 DM and has been on insulin pump therapy for at least 3 months prior to signature of the informed consent
* patients use CGM component as part as part of the continuous subcutaneous insulin infusion (CSII) therapy for a minimum of 1 month

Exclusion Criteria:

* participation in any other trial
* any disease or drug treatment that can interfere with the outcome of sensor usage
* using CGM in CSII < 3 days/week
* patients not willing to sign informed consent
* abuse of alcohol or drugs (exception of nicotine consumption)
* eating disorder, anorexia, bulimia or other mental disorders

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diabetes mellitus, type 1
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tsioli C, Danne T für die RANSuP-Studiengruppe. RANSuP-Registerstudie: Anwendung der Sensorunterstützten Pumpentherapie unter Alltagsbedingungen. Diabetologie und Stoffwechsel 2013; 8: S62

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group
Started | 75
Completed | 67
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Group
Number analyzed (Participants) | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 55
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.88 (16.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 39
Region of Enrollment [Number; unit: participants]
  Germany | 75

OUTCOME MEASURES:

1. Primary Outcome: Number (n) of Excursions <70 mg/dl Per Sensor Day at Baseline and 3 Months
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: excursions
Arm/Group | Intervention Group
Number analyzed (Participants) | 67
excursions
  Baseline | 1.26 (0.69)
  3 months | 0.98 (0.59)
Statistical Analysis 1: Comparison: Intervention Group; Test type: Other; p = 0.001, t-test, 2 sided

2. Secondary Outcome: Number (n) of Excursions <40 mg/dl Per Sensor Day at Baseline and 3 Months
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: excursions
Arm/Group | Intervention Group
Number analyzed (Participants) | 67
excursions
  Baseline | 0.19 (0.22)
  3 months | 0.16 (0.21)
Statistical Analysis 1: Comparison: Intervention Group; Test type: Other; p = 0.12, Wilcoxon Signed-Rank Test

3. Secondary Outcome: Hemoglobin A1c (HbA1c) Values (%) at Baseline and 3 Months
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- Intervention Group: Patients treated with Sensor-augmented pump therapy with insulin pump Paradigm VEO® and use continuous glucose monitoring (CGM).
Arm/Group | Intervention Group
Number analyzed (Participants) | 67
Percentage
  Baseline | 7.96 (0.93)
  3 months | 7.90 (0.97)
Statistical Analysis 1: Comparison: Intervention Group; Test type: Other; p = 0.30, Wilcoxon Signed-Rank Test

4. Secondary Outcome: Interstitial Sensor Glucose Concentration (mg/dl) at Baseline and 3 Months
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Intervention Group
Number analyzed (Participants) | 67
mg/dl
  Baseline | 154.80 (24.21)
  3 months | 159.06 (25.78)
Statistical Analysis 1: Comparison: Intervention Group; Test type: Other; p = 0.03, t-test, 2 sided

5. Secondary Outcome: Sensor Wearing Time (Sensor Days/Calendar Week) at Baseline and 3 Months
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: sensor days/calendar week
Groups:
- Intervention Group: Patients treated with sensor augmented pump (SAP) therapy with insulin pump Paradigm VEO® and use continuous glucose monitoring (CGM).
  sensor augmented pump (SaP)
Arm/Group | Intervention Group
Number analyzed (Participants) | 67
sensor days/calendar week
  Baseline | 5.6 (1.0)
  3 months | 5.01 (1.46)
Statistical Analysis 1: Comparison: Intervention Group; Test type: Other; p = 0.04, Wilcoxon Signed-Rank Test

6. Secondary Outcome: Area Under the Curve (AUC) in Hypoglycemic Region (< 70mg/dl) at Baseline and 3 Months
Description: Area under the curve (AUC) in hypoglycemic region (< 70mg/dl) at baseline (1 month before the start of the study) and 3 months during the study.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mg/dl*day
Arm/Group | Intervention Group
Number analyzed (Participants) | 67
mg/dl*day
  Baseline | 0.07 (0.35)
  3 months | 0.028 (0.026)
Statistical Analysis 1: Comparison: Intervention Group; Test type: Other; p = 0.35, Wilcoxon Signed-Rank Test

7. Secondary Outcome: Area Under the Curve (AUC) in Hyperglycemic Region (>140mg/dl) at Baseline and 3 Months
Description: Area under the curve (AUC) in hyperglycemic region (>140mg/dl) at baseline (1 month before the start of the study) and 3 months during the study.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mg/dl*day
Arm/Group | Intervention Group
Number analyzed (Participants) | 67
mg/dl*day
  Baseline | 1.32 (0.87)
  3 months | 1.79 (1.44)
Statistical Analysis 1: Comparison: Intervention Group; Test type: Other; p = 0.001, Wilcoxon Signed-Rank Test

8. Secondary Outcome: Time in Hyperglycemic Region Per Sensor Day at Baseline and 3 Months
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: min/sensor day
Arm/Group | Intervention Group
Number analyzed (Participants) | 67
min/sensor day
  Baseline | 737.62 (232.56)
  3 months | 771.00 (426.52)
Statistical Analysis 1: Comparison: Intervention Group; Test type: Other; p = 0.61, Wilcoxon Signed-Rank Test

9. Secondary Outcome: Number of Automatic Low Glucose Suspend (LGS) Activations in Daytime (6:00 - 22:00 Hrs) at Baseline and 3 Months
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: activations/patient/sensor day
Arm/Group | Intervention Group
Number analyzed (Participants) | 67
activations/patient/sensor day
  Baseline | 0.62 (0.71)
  3 months | 0.73 (0.83)
Statistical Analysis 1: Comparison: Intervention Group; Test type: Other; p = 0.1, Wilcoxon Signed-Rank Test

10. Secondary Outcome: Number of Automatic Low Glucose Suspend (LGS) Activations in Nighttime (22:00 - 6:00 Hrs) at Baseline and 3 Months
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: activations/patient/sensor day
Arm/Group | Intervention Group
Number analyzed (Participants) | 67
activations/patient/sensor day
  Baseline | 0.22 (0.29)
  3 months | 0.25 (0.29)
Statistical Analysis 1: Comparison: Intervention Group; Test type: Other; p = 0.22, Wilcoxon Signed-Rank Test

11. Secondary Outcome: Interstitial Sensor Glucose Excursions After Meals (Amplitude of Excursions) at Baseline and 3 Months
Time Frame: Baseline and 3 months
Population: Meals were not adequately documented, so that a meaningful analysis was not possible
Arm/Group | Intervention Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No